CLINICAL TRIAL: NCT03537313
Title: Vaginal Douching and Painting in Women Who Underwent Total Abdominal Hysterectomy: A Factorial 2-by-2 Open-labeled Randomized Controlled Trial
Brief Title: Vaginal Douching and Painting in Women Who Underwent Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: RJVAG001
Record Dates: First submitted 2018-05-11; First posted 2018-05-25 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2018-05

CONDITIONS: Febrile Morbidity

STUDY DESIGN:
Intervention Model Description: Factorial 2-by-2 open labeled randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control-douching group (No Intervention): No preoperative vagina douching
- Control-painting group (No Intervention): No intra-operative vagina painting
- Vaginal douching group (Experimental): Preoperative vaginal douches with povidone-iodine solution
  Interventions: Procedure: Vagina douching
- Vaginal painting group (Experimental): Intra-operative vaginal painting with povidone-iodine solution
  Interventions: Procedure: Vagina painting

INTERVENTIONS:
Procedure: Vagina douching — Vaginal douches with 1000 ml of 1% povidone-iodine solution on the night before surgery and again on the morning of surgery
  Arms: Vaginal douching group
Procedure: Vagina painting — Vaginal painting of vagina stump after hysterectomy with 10% povidone-iodine solution 30 ml
  Arms: Vaginal painting group

SUMMARY:
Comparison of the effectiveness of povidone-iodine douching and painting for reducing febrile morbidity after total abdominal hysterectomy

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is the most common gynecologic operation worldwide. The two most common complications after TAH are febrile and infectious morbidities, incidence varying between 5 and 50 percent. After performing TAH, vaginal canal must be breached and closed to be blind-pouch stump. Routing vaginal douching at the night before and on the morning of the surgical date, and intra-operative painting are routinely practiced. However, no good quality of evidence base supports the effectiveness of vaginal douching and painting in preventing febrile and infectious morbidities after TAH.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergoing total abdominal hysterectomy
* Woman who agrees to participate in this study

Exclusion Criteria:

* Women with history of sea-food or iodine allergy
* Women who undergo emergency TAH
* Women who have intestinal resection in this operation
* Women who have active pelvic inflammatory disease before operation
* Women who have fever before operation
* Women who received antibiotic within 1 weeks before operation
* Women who be immunocompromised host

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Febrile morbidity | Day 1-7 after surgery
  Defined as the presence of an oral temperature > 38 o C (100.4 o F) on two occasions at least 4 hours apart in the post-operative period excluding the first 24 hours

SECONDARY OUTCOMES:
Vaginal cuff infection | 2 weeks after surgery
  Defined as redness, tenderness, infiltration or abscess at vaginal cuff
Other infectious morbidities | 2 weeks after surgery
  Defined by the presence of a urinary tract infection, abdominal wound infection, or pneumonitis; urinary tract infection defined as symptomatic infection with a mid-steam urine specimen showed bacterial growth > 105 bacteria/ml of urine; surgical wound infection defined as redness, tenderness, infiltration or abscess; pneumonitis defined as fever, physical and radiological findings of consolidation

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand